CLINICAL TRIAL: NCT05645861
Title: MAnagement of Systolic Blood Pressure During Thrombectomy by Endovascular Route for Acute Ischaemic STROKE: the MASTERSTROKE Trial
Brief Title: MAnagement of Systolic Blood Pressure During Thrombectomy by Endovascular Route for Acute Ischaemic STROKE
Acronym: MASTERSTROKE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Auckland City Hospital (Other Government)
Collaborators: The Australian and New Zealand College of Anaesthetists (ANZCA) (Unknown); Neurological Foundation of New Zealand (Unknown); The University of Queensland (Other); Auckland Medical Research Foundation (Other); Auckland Hospitals Research and Endowment Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MasterStroke vs 1.4; 1920 PG (Other Grant/Funding Number: Neurological Foundation); 22/001 (Other Grant/Funding Number: Australia New Zealand College of Anaesthesia); A+ 8173 (Other Grant/Funding Number: Auckland Hospitals Research and Endowment Fund); 2119013 (Other Grant/Funding Number: Auckland Medical Research Foundation); ACTRN12619001274167 (Registry Identifier: Australia New Zealand Clinical Trials Registry)
Record Dates: First submitted 2022-11-30; First posted 2022-12-12 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-11

CONDITIONS: Stroke; Embolus Cerebral; Blood Pressure
MeSH Terms: conditions — Stroke; Intracranial Embolism

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant, investigators and outcome assessors are blinded to randomization allocation using opaque envelopes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Augmented - Systolic Blood Pressure (SBP) at 170mmHg +/- 10 mmHg (Active Comparator): Techniques used to target SBP will not be controlled for and will be at the discretion of the procedural anaesthetist to manage blood pressure, this can include vasopressors, intravenous fluids, titration of anaesthetic maintenance drugs and use of other vasoactive drugs.
  Interventions: Procedure: Blood pressure management of Systolic Blood Pressure to maintain target range +/- 10 mmHg
- Standard - Systolic Blood Pressure (SBP) at 140mmHg +/- 10 mmHg (Active Comparator): Techniques used to target SBP will not be controlled for and will be at the discretion of the procedural anaesthetist to manage blood pressure, this can include vasopressors, intravenous fluids, titration of anaesthetic maintenance drugs and use of other vasoactive drugs.
  Interventions: Procedure: Blood pressure management of Systolic Blood Pressure to maintain target range +/- 10 mmHg

INTERVENTIONS:
Procedure: Blood pressure management of Systolic Blood Pressure to maintain target range +/- 10 mmHg — Techniques used to target SBP will not be controlled for and will be at the discretion of the procedural anaesthetist to manage blood pressure, this can include vasopressors, intravenous fluids, titration of anaesthetic maintenance drugs and use of other vasoactive drugs.

SUMMARY:
Stroke is the third most common cause of death in New Zealand and is one of the leading causes of long-term disability at all ages. A life-saving clot retrieval procedure can save lives and prevent disability of patients with ischaemic stroke who get to hospital in time. In New Zealand, 90% of clot retrieval procedures are performed under general anaesthesia. Many anaesthetic drugs can affect blood pressure (BP) and blood flow within the brain. Increasing BP during the procedure could provide additional benefits in this devastating disease. A large trial is needed to investigate BP management during clot retrieval.

DETAILED DESCRIPTION:
Internationally stroke ranks second among all causes of disability and is adding to considerable worldwide healthcare burden. Over the last 5 years a new procedure to remove clots (Endovascular Thrombectomy - EVT) has been effective for the treatment of acute large strokes, with significant reductions in long term patient disability compared to standard treatment. However, there minimal guidance on blood pressure management during the procedure. The brain is especially vulnerable to low blood pressure during the acute stroke period due to low blood supply, impairment of how the brain regulates blood flow and further falls in blood flow to the brain. High blood pressure may be beneficial due to increased blood flow in areas at risk during this time. It could be harmful due to brain injury process, swelling, and bleeding into the brain. Conversely, relatively low blood pressure could be harmful. Current evidence is limited to large observational studies. This randomised controlled study will examine the safety and efficacy of two systolic blood pressures (SBP) management arms during general anaesthesia for EVT on outcomes in patients with acute ischaemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with anterior circulation stroke (ICA or proximal M1 or M2 segment of MCA) treated with ECR within 6 hrs of stroke onset and ECR patients presenting within 6-24 hours and favourable penumbra on perfusion scanning (see criteria 1-3).

Additional criteria in the 6 to 24-hour window.

1. 'wake up' stroke; CT with no (or at most minimal) acute infarction or
2. patient 80 years or older (NIHSS of 10 and infarct volume less than 21 ml on DWI or CT perfusion-CBF)
3. patient less than 80 years (NIHSS of 10 and infarct volume less than 31 ml on DWI or CT perfusion-CBF NIHSS of 20 and infarct volume less than 51 ml on DWI or CT perfusion-CBF).

Exclusion Criteria:

* Rescue"' procedures eg acute ischaemic stroke associated with major medical procedures such as coronary artery stenting and coronary artery bypass

  * pre-stroke mRS>=3
  * not having GA
  * terminal illness with expected survival <1 year
  * pregnancy
  * cardiovascular conditions where BP targeting will be contra-indicated
  * unable to participate in 3-month follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2019-11-28 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Day 90 Modified Rankin Score | 90 days Post Thrombectomy
  The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 (no symptoms at all) to 5 (severe disability). A separate category of 6 is usually added for patients who are deceased.

SECONDARY OUTCOMES:
Independent functionality | 90 days Post Thrombectomy
  Independent functional outcome as determined by a modified Rankin Score of 0,1,or 2 at 90 Days. The Modified Rankin Score (mRS) is a 6 point disability scale with possible scores ranging from 0 (no symptoms at all) to 5 (severe disability). A separate category of 6 is usually added for patients who are deceased.
Days Alive out of Hospital (DAOH) | 90 days Post Thrombectomy
  The number of days a participant spends at home in the first 90 days post-stroke (home days/DAH90 confirmed by patient follow-up and clinical note review.
All cause mortality | 90 days Post Thrombectomy
  All cause mortality confirmed by patient follow-up and clinical note review.
Intraprocedural complications | From randomisation until 36 hours post treatment
  Proportion of patients with intra-procedural complications (target vessel dissection, intracerebral haemorrhage, groin haematoma) as documented in medical records.
Complicaiton of importance - symptomatic intracranial haemorrhage | From randomisation until 36 hours post treatment
  Proportion of patients with symptomatic intracranial haemorrhage (within 36 hours of treatment) as documented in medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Doug Campbell, Dr, Principal Investigator — Auckland City Hospital
Locations (6):
- Australia (3):
  - Royal North Shore Hospital, Sydney, New South Wales
  - Gold Coast University Hospital, Southport, Queensland
  - Metro South Hospital and Health Service via the Princess Alexandra Hospital, Woolloongabba, Queensland
- New Zealand (3):
  - Auckland City Hopsital, Auckland, Auckland
  - Christchurch Hospital, Christchurch, Canterbury
  - Wellington Regional Hospital, Newton, Wellington Region

IPD SHARING:
Plan to Share IPD: No
At this time the steering committee have not developed an IPD data sharing plan. Once the decision has been made regarding this process the information will be updated accordingly.

REFERENCES:
- See also: Australia New Zealand College of Anaesthesia current research — https://www.anzca.edu.au/profiles/ctn-trials/underway/masterstroke-trial

DOCUMENTS (2):
  • Study Protocol (2024-08-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT05645861/Prot_001.pdf
  • Statistical Analysis Plan (2025-11-17): https://cdn.clinicaltrials.gov/large-docs/61/NCT05645861/SAP_002.pdf